CLINICAL TRIAL: NCT05700565
Title: Treatment of Immune-related Adverse Events Refractory to Standard Therapy and Associated Changes in Immunophenotype
Acronym: PRIA
Status: Recruiting | Type: Observational
Sponsor: Lucie Heinzerling (Other)
Responsible Party: Sponsor-Investigator, Lucie Heinzerling, Prof. Dr. (MPH), LMU Klinikum
Organization: LMU Klinikum (Other)
Other Study IDs: LMUKlinikum
Record Dates: First submitted 2022-11-04; First posted 2023-01-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Immune-related Adverse Event
Keywords: Steroid-refractory; Steroid-dependent
MeSH Terms: interventions — Photopheresis; Immunomodulating Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (Serum, EDTA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Steroid-refractory or dependent immune-related adverse events: Immune-related adverse events (irAE) after immune checkpoint inhibitor therapy (PD-1/PD-L1 or PD-1 + CTLA4 blockade) refractory to therapy with corticosteroids or inability to taper corticosteroids to prednisone equivalent <= 5mg
  Interventions: Other: Extracorporeal photopheresis; Other: Other immunosuppressive or immunomodulatory drugs

INTERVENTIONS:
Other: Extracorporeal photopheresis — ECP consists of the three steps of leukapheresis, photoactivation and reinfusion and has immunomodulatory effects (modulation of dendritic cells, change in cytokine profile, induction of T cell subpopulations). Indications are currently the treatment of Sézary syndrome, Graft-versus-host disease (GvHD), organ transplant rejection and systemic scleroderma.
Other: Other immunosuppressive or immunomodulatory drugs — Other immunosuppressive or immunomodulatory drugs

SUMMARY:
This study is an open, monocentric study. It includes patients with irAE refractory to standard therapy or patients where corticosteroids cannot be tapered. Patients will either be treated with ECP or second line immunosuppressive therapy according to investigator's choice. Patients will be followed for 24 weeks after first treatment.

DETAILED DESCRIPTION:
At inclusion patient history including type of tumor and immunotherapy will be obtained.

At all visits symptoms, changes in concomitant medication, a medical assessment and laboratory investigations will be performed. Blood sampling for safety analysis and for investigating the immunophenotype will be performed at baseline, week 1, 4, 8 and 12.

Laboratory values assessed include:

* Complete blood count
* Chemistry including liver enzymes (AST, ALT) and total bilirubin in the case of immune-related hepatitis, CK in case of myositis, creatinine in case of nephritis
* Inflammatory markers: CRP, IL-6, Procalcitonin Peripheral blood mononuclear cells (PBMC) will be used to determine immunophenotype, including the amount of NK-cells, regulatory T- cells and myeloid-derived suppressor cells (MDSC) as well as the expression of inflammatory markers. Biological samples will be frozen for later analysis.

Additionally, patients will assess their symptoms and their quality of life by a self-administered questionnaire at baseline and week 4, 8 and 12. Quality of life will be assessed by EORTC QLQ-C30. All irAE will be graded according to CTCAE.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must we willing and able to comply with scheduled visits and must have given written informed consent.
2. irAE after immune checkpoint inhibitor therapy (PD-1/PD-L1 or PD-1 + CTLA4 blockade)
3. irAE refractory to therapy with corticosteroids or inability to taper corticosteroids to prednisone equivalent <= 5mg. An irAE is defined as refractory if corticosteroids do not improve symptoms within 72 hours. The inability to taper corticosteroids is defined as relapse on standard tapering of 1 mg/kg corticosteroid over 28 days.

Exclusion Criteria:

1. Contraindications for the treatment with ECP including a known sensitivity to psoralen compounds such as 8-MOP, comorbidities that may result in photosensitivity, aphakia, history of heparin-induced thrombocytopenia, unsatisfactory cardio-circulatory function, low hematocrit values
2. Pregnancy
3. Body weight less than 40 kg.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with irAE after immune checkpoint inhibitor therapy (PD-1/PD-L1 or PD-1 + CTLA4 blockade) refractory to therapy with corticosteroids or inability to taper corticosteroids to prednisone equivalent <= 5mg. An irAE is defined as refractory if corticosteroids do not improve symptoms within 72 hours. The inability to taper corticosteroids is defined as relapse on standard tapering of 1 mg/kg corticosteroid over 28 days.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Immunophenotype | 12 weeks
  Characterisation of peripheral mononuclear blood cells

SECONDARY OUTCOMES:
Developement of grade of irAE | 12 weeks
  irAE symptoms graded according to CTCAE v5.0
Patient quality of life | 12 weeks
  Quality of life assessed by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Heinzerling, Principal Investigator — Department of Dermatology and Allergy, University Hospital, LMU Munich
Locations (1):
- LMU Klinikum Hauttumorzentrum, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ertl C, Ruf T, Hammann L, Piseddu I, Wang Y, Schmitt C, Garza Vazquez X, Kabakci C, Bonczkowitz P, de Toni EN, David-Rus R, Srour J, Tomsitz D, French LE, Heinzerling L. Extracorporeal photopheresis vs. systemic immunosuppression for immune-related adverse events: Interim analysis of a prospective two-arm study. Eur J Cancer. 2024 Nov;212:115049. doi: 10.1016/j.ejca.2024.115049. Epub 2024 Sep 27. PMID 39383612